CLINICAL TRIAL: NCT04084756
Title: Couples Intervention to Improve Mental Health
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Wesleyan University (Other)
Collaborators: University of Utah (Other); Military Suicide Research Consortium (Other)
Responsible Party: Principal Investigator, Alexis May, Assistant Professor, Wesleyan University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 00113793; W81XWH-16-2-0004 (Other Grant/Funding Number: Military Suicide Research Consortium)
Record Dates: First submitted 2019-09-03; First posted 2019-09-10 (Actual); Last update posted 2022-05-12 (Actual); Status verified 2022-05

CONDITIONS: Suicide
MeSH Terms: conditions — Suicide

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Couples Crisis Response Plan (Experimental)
  Interventions: Behavioral: Couples Crisis Response Plan
- Mental Health Education (Active Comparator)
  Interventions: Behavioral: Mental Health Education

INTERVENTIONS:
Behavioral: Couples Crisis Response Plan — The CCRP is a single session therapist-facilitated suicide prevention intervention conducted with a dyad
  Arms: Couples Crisis Response Plan
Behavioral: Mental Health Education — The Mental Health Education session is a single session therapist-facilitated mental health psychoeducation session conducted with a dyad
  Arms: Mental Health Education

SUMMARY:
Over the last decade, suicide rates have risen within the military and have remained high. Converging evidence suggests that suicide prevention efforts may be enhanced by explicitly including family members in treatment. The study's objectives are to test the effect of the CCRP, a targeted single session couples intervention on suicide ideation among military service members and Veterans, and to understand how the use of the CCRP impacts suicide risk during the 6 months immediately postdischarge from a psychiatric inpatient unit.

DETAILED DESCRIPTION:
Over the last decade, suicide rates have risen within the military and have remained high. Converging evidence suggests that suicide prevention efforts may be enhanced by explicitly including family members in treatment, however no couple-bases suicide-specific interventions exist.

The study's objectives are to test the effect of the Couples Crisis Response Plan (CCRP), a targeted single-session couples intervention, on suicide ideation among military service members and Veterans, and to understand how the use of the CCRP impacts suicide risk during the period of time immediately post-discharge from a psychiatric inpatient unit. The CCRP will be compared to an active control condition (mental health education).

The primary aim is to compare the effect of the CCRP to an active control condition on suicide ideation in the 6 months following treatment among military service members and Veterans who have been psychiatrically hospitalized for acute suicide risk and their partners. The CCRP is specifically adapted for use with partnered service members at elevated risk for suicide. A secondary aim is to determine how use of the CCRP skills impacts suicidal ideation over time and identify the role partners play in encouraging use of the plan and managing suicide risk.

ELIGIBILITY:
Inclusion Criteria:

1. military service member (active duty or veteran) of any branch or component that has served since 9/11/2001 or the partner of such a service member;
2. that the service member reports active suicide ideation and/or a suicide attempt within the previous 30 days;
3. that the service member is in a committed, exclusive, cohabiting relationship of at least 6 months;
4. the willingness of the service member's partner to participate in research.

Exclusion Criteria:

1. a psychiatric condition, medical condition, or cognitive disability/deficit that precludes the ability of either partner to provide informed consent
2. physical aggression within the past year reported by either partner on a behaviorally-anchored screener for moderate to severe partner violence or extreme relationship distress (a score of of less than 9 on the Couples Satisfaction Index-4)
3. inability of either partner to read or speak English

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2019-08-01 (Actual); Primary Completion 2022-09 (Estimated); Study Completion 2022-09 (Estimated)

PRIMARY OUTCOMES:
Change in suicidal thoughts and behaviors since baseline measured by the Scale for Suicidal Ideation | Assessed at baseline and 1, 3 and 6-months follow ups
  Self-report assessment of severity of suicidal thoughts and behaviors. Items 1-19 are summed (range: 0-38) and higher scores indicate greater suicide severity. Measured at baseline, hospital discharge, and 1, 3, and 6 month follow ups.

SECONDARY OUTCOMES:
Change in number of suicide attempts from baseline | Assessed at baseline and 1, 3 and 6-months follow ups
  The change in number of suicide attempts from baseline will be assessed through participants' responses to the Self-Injurious Thoughts and Behaviors Interview. The Self-Injurious Thoughts and Behaviors Interview is a structured interview assessing history of suicidal thoughts and behaviors, including suicide attempt history (dates, methods, and severity (e.g., need for medical attention) of previous suicide attempts). An increased number of suicide attempts at any assessment is considered a worse outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Alexis May, PhD, Principal Investigator — Wesleyan Univerity; Craig Bryan, PsyD, APBB, Principal Investigator — University of Utah
Locations (1):
- Salt Lake Behavioral Health, Salt Lake City, Utah, United States